CLINICAL TRIAL: NCT01708629
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Induction and Maintenance Regimens of Brodalumab Compared With Placebo and Ustekinumab in Subjects With Moderate to Severe Plaque Psoriasis: AMAGINE-3
Brief Title: Efficacy and Safety of Brodalumab Compared With Placebo and Ustekinumab in Moderate to Severe Plaque Psoriasis Subjects
Acronym: AMAGINE-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120104
Record Dates: First submitted 2012-09-21; First posted 2012-10-17 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Plaque Psoriasis
Keywords: psoriasis, brodalumab, AMG 827
MeSH Terms: conditions — Psoriasis | interventions — brodalumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 210 mg brodalumab (Experimental): Administered by subcutaneous (SC) injection until week 12. At week 12, participants are rerandomized to schedule 1, 2, 3, or 4.
  Interventions: Drug: 210 mg brodalumab
- 140 mg brodalumab (Experimental): Administered by subcutaneous (SC) injection until week 12. At week 12, participants are rerandomized to schedule 1, 2, 3, or 4.
  Interventions: Drug: 140 mg brodalumab
- ustekinumab (Active Comparator): Administered by subcutaneous (SC) injection per the labeled dosing regimen.
  Interventions: Drug: ustekinumab
- Placebo (Placebo Comparator): Administered by SC injection until week 12. At week 12 participants are assigned to 210 mg brodalumab.
  Interventions: Drug: 210 mg brodalumab; Drug: placebo

INTERVENTIONS:
Drug: 210 mg brodalumab — 210 mg brodalumab administered SC
  Other Names: Siliq
  Arms: 210 mg brodalumab; Placebo
Drug: 140 mg brodalumab — 140 mg brodalumab administered SC
  Other Names: Siliq
  Arms: 140 mg brodalumab
Drug: ustekinumab — 45 mg or 90 mg ustekinumab administered SC per the labeled dosing regimen.
  Other Names: Stelara
  Arms: ustekinumab
Drug: placebo — placebo administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of brodalumab at two different doses compared with placebo in participants with moderate to severe plaque psoriasis.

A second purpose of this study is to assess the safety and efficacy brodalumab at two different doses compared with ustekinumab in participants with moderate to severe plaque psoriasis.

A third purpose of this study is to assess the safety and efficacy of 4 maintenance regimens of brodalumab.

DETAILED DESCRIPTION:
This study assess the safety and efficacy of brodalumab at two different doses compared with placebo in participants with moderate to severe plaque psoriasis.

A second purpose of this study is to assess the safety and efficacy brodalumab at two different doses compared with ustekinumab in participants with moderate to severe plaque psoriasis.

A third purpose of this study is to assess the safety and efficacy of 4 maintenance regimens of brodalumab.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had stable moderate to severe plaque psoriasis for at least 6 months
* Subject has involved body surface area (BSA) ≥ 10%, PASI ≥ 12, and sPGA ≥ 3 at screening and at baseline

Exclusion Criteria:

* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions at (eg, eczema) that would interfere with study evaluations
* Subject has known history of Crohn's disease
* Subject has any other significant concurrent medical condition or laboratory abnormalities, as defined in the study protocol
* Subject has not stopped using certain psoriasis therapies as defined in the study protocol
* Subject has previously used ustekinumab or any anti-IL-17 biologic therapy
* Subject is pregnant or breastfeeding, or planning to become pregnant while enrolled in the study
* Female subject is unwilling to use highly effective methods of birth control unless 2 years post-menopausal or surgically sterile

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1881 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (138):
- United States (69):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, Encino, California
  - Research Site, Fremont, California
  - Research Site, Fullerton, California
  - Research Site, Irvine, California
  - Research Site, Los Angeles, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Denver, Colorado
  - Research Site, Farmington, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Alpharetta, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Arlington Heights, Illinois
  - Research Site, Champaign, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Wheaton, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, New Albany, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Clarkston, Michigan
  - Research Site, Clinton Township, Michigan
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, East Windsor, New Jersey
  - Research Site, Hoboken, New Jersey
  - Research Site, Verona, New Jersey
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, High Point, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Lake Oswego, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Exton, Pennsylvania
  - Research Site, Johnston, Rhode Island
  - Research Site, Greer, South Carolina
  - Research Site, Bartlett, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Bellaire, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Webster, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Clarksburg, West Virginia
- Australia (8):
  - Research Site, Camperdown, New South Wales
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Hectorville, South Australia
  - Research Site, Fremantle, Western Australia
- Belgium (7):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Montigny-le-Tilleul
- Canada (13):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Richmond Hill, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Drummondville, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Hyacinthe, Quebec
- France (7):
  - Research Site, Créteil
  - Research Site, Limoges
  - Research Site, Nice
  - Research Site, Poitiers
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Greece (6):
  - Research Site, Chaïdári, Athens
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Marousi
  - Research Site, Thessaloniki
- Hungary (6):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Szeged
  - Research Site, Szolnok
  - Research Site, Szombathely
- Italy (4):
  - Research Site, Bologna
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Roma
- Latvia (2):
  - Research Site, Riga
  - Research Site, Ventspils
- Poland (12):
  - Research Site, Bialystok
  - Research Site, Dąbrówka
  - Research Site, Gdansk
  - Research Site, Iwonicz-Zdrój
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Stalowa Wola
  - Research Site, Świdnik
  - Research Site, Warsaw
- Russia (4):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lebwohl MG, Armstrong AW, Alexis AF, Lain EL, Jacobson AA. Efficacy of Brodalumab in Patients with Psoriasis and Risk Factors for Treatment Failure: A Review of Post Hoc Analyses. Dermatol Ther (Heidelb). 2024 Oct;14(10):2709-2726. doi: 10.1007/s13555-024-01264-3. Epub 2024 Sep 12. PMID 39264399
- [Derived] Kokolakis G, Vadstrup K, Hansen JB, Carrascosa JM. Increased Skin Clearance and Quality of Life Improvement with Brodalumab Compared with Ustekinumab in Psoriasis Patients with Aggravating Lifestyle Factors. Dermatol Ther (Heidelb). 2021 Dec;11(6):2027-2042. doi: 10.1007/s13555-021-00618-5. Epub 2021 Oct 2. PMID 34606048
- [Derived] Gottlieb A, Lebwohl M, Liu C, Israel RJ, Jacobson A. Malignancy Rates in Brodalumab Clinical Studies for Psoriasis. Am J Clin Dermatol. 2020 Jun;21(3):421-430. doi: 10.1007/s40257-020-00512-4. PMID 32207067
- [Derived] McMichael A, Desai SR, Qureshi A, Rastogi S, Alexis AF. Efficacy and Safety of Brodalumab in Patients with Moderate-to-Severe Plaque Psoriasis and Skin of Color: Results from the Pooled AMAGINE-2/-3 Randomized Trials. Am J Clin Dermatol. 2019 Apr;20(2):267-276. doi: 10.1007/s40257-018-0408-z. PMID 30471012
- [Derived] Langley RG, Armstrong AW, Lebwohl MG, Blauvelt A, Hsu S, Tyring S, Rastogi S, Pillai R, Israel R. Efficacy and safety of brodalumab in patients with psoriasis who had inadequate responses to ustekinumab: subgroup analysis of two randomized phase III trials. Br J Dermatol. 2019 Feb;180(2):306-314. doi: 10.1111/bjd.17318. Epub 2018 Dec 27. PMID 30328108
- [Derived] Lebwohl M, Strober B, Menter A, Gordon K, Weglowska J, Puig L, Papp K, Spelman L, Toth D, Kerdel F, Armstrong AW, Stingl G, Kimball AB, Bachelez H, Wu JJ, Crowley J, Langley RG, Blicharski T, Paul C, Lacour JP, Tyring S, Kircik L, Chimenti S, Callis Duffin K, Bagel J, Koo J, Aras G, Li J, Song W, Milmont CE, Shi Y, Erondu N, Klekotka P, Kotzin B, Nirula A. Phase 3 Studies Comparing Brodalumab with Ustekinumab in Psoriasis. N Engl J Med. 2015 Oct;373(14):1318-28. doi: 10.1056/NEJMoa1503824. PMID 26422722
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Ustekinumab | Placebo
Started | 624 | 629 | 313 | 315
Completed | 608 | 604 | 303 | 301
Not Completed | 16 | 25 | 10 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Ustekinumab | Placebo | Total
Number analyzed (Participants) | 624 | 629 | 313 | 315 | 1881
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 578 | 589 | 292 | 300 | 1759
  >=65 years | 46 | 40 | 21 | 15 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (13.3) | 44.6 (13.0) | 44.8 (13.1) | 44.2 (12.5) | 44.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193 | 192 | 101 | 107 | 593
  Male | 431 | 437 | 212 | 208 | 1288
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 1 | 0 | 7
  Asian | 20 | 27 | 12 | 9 | 68
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 1 | 1 | 8
  Black or African American | 17 | 22 | 13 | 6 | 58
  White | 565 | 569 | 280 | 294 | 1708
  More than one race | 2 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 14 | 4 | 6 | 5 | 29
Region of Enrollment [Number; unit: participants]
  Greece | 21 | 23 | 11 | 10 | 65
  Canada | 72 | 75 | 38 | 34 | 219
  Latvia | 33 | 32 | 15 | 16 | 96
  Russia | 23 | 21 | 9 | 12 | 65
  Hungary | 17 | 16 | 10 | 7 | 50
  Belgium | 8 | 8 | 3 | 6 | 24
  United States | 276 | 278 | 140 | 141 | 835
  Poland | 127 | 128 | 63 | 63 | 381
  Italy | 2 | 3 | 1 | 2 | 8
  Australia | 17 | 16 | 9 | 8 | 50
  France | 28 | 29 | 14 | 16 | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Psoriasis Area Severity Index (PASI) 75 at Week 12
Description: The Psoriasis Area and Severity Index Score is used as a scale to show change from Baseline of study to a certain point. PASI Score ranges from (0) no disease to (72) maximal disease. The proportion of subjects achieving 75% improvement in Psoriasis Area and Severity Index, PASI75, was assessed.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Ustekinumab: Administered by subcutaneous (SC) injection until week 12. Participants using Ustekinumab were not rerandomized at week 12, and continued to receive ustekinumab.
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo | Ustekinumab
Number analyzed (Participants) | 624 | 629 | 315 | 313
Participants | 531 | 435 | 19 | 217

2. Primary Outcome: Percentage of Participants With Static Physician Global Assessment (sPGA) Success Score (Score of 0 or 1) at Week 12 - Comparison to Placebo
Description: Static Physician Global Assessment (sPGA) measures the physician's impression of the disease. Possible scores are (0 [clear] to 5 [severe]). Success was defined by a score of 0 or 1 (clear to almost clear).
Time Frame: 12 weeks
Population: sPGA was only assessed as a comparison of Brodalumab (210mg and 140mg) to Placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo
Number analyzed (Participants) | 624 | 629 | 315
Participants | 497 | 377 | 13

ADVERSE EVENTS:
Groups:
- Ustekinumab: Administered by subcutaneous (SC) injection until week 12. At week 12, participants are rerandomized to schedule 1, 2, 3, or 4.
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo | Ustekinumab
Serious Adverse Events (participants affected / at risk) | 9/624 | 10/629 | 3/315 | 2/313
Other Adverse Events (participants affected / at risk) | 353/624 | 329/629 | 152/315 | 168/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 210 mg Brodalumab (N=624) | 140 mg Brodalumab (N=629) | Placebo (N=315) | Ustekinumab (N=313)
Gastroenteritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Altered State of Consciousness (General disorders) | 1 | 0 | 0 | 0
Appendicitus (Immune system disorders) | 0 | 1 | 0 | 0
Arthritis (General disorders) | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Bladder Cancer (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Cerebrovascular Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cholecystitis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Diverticulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Encephalopathy (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Erythrodermic Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 1 | 0 | 0 | 0
Meningitis Cryptoccocal (Infections and infestations) | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Nervous system disorders) | 0 | 1 | 0 | 0
Overdose (General disorders) | 1 | 0 | 0 | 0
Peritonsillar Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 210 mg Brodalumab (N=624) | 140 mg Brodalumab (N=629) | Placebo (N=315) | Ustekinumab (N=313)
Nasopharyngitis (Infections and infestations) | 31 | 36 | 22 | 16
Upper respiratory tract Infection (Infections and infestations) | 33 | 19 | 17 | 16
Urinary Tract Infection (Infections and infestations) | 11 | 5 | 3 | 8
Pharyngitis (Infections and infestations) | 9 | 5 | 6 | 4
Influenza (Infections and infestations) | 8 | 5 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 25 | 6 | 10
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 10 | 11 | 3 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 11 | 5 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 9 | 2 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 7 | 7 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 17 | 15 | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 6 | 9 | 9 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 4 | 6 | 1 | 0
Fatigue (General disorders) | 20 | 20 | 6 | 4
Influenza Like Illness (General disorders) | 6 | 7 | 3 | 1
Pyrexia (General disorders) | 6 | 4 | 3 | 3
Injection Site Pain (General disorders) | 4 | 1 | 2 | 4
headache (Nervous system disorders) | 21 | 32 | 14 | 11
Dizziness (Nervous system disorders) | 7 | 3 | 1 | 1
Sciatica (Nervous system disorders) | 3 | 4 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 14 | 6 | 4 | 3
Nausea (Gastrointestinal disorders) | 11 | 11 | 2 | 1
Toothache (Gastrointestinal disorders) | 7 | 4 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 14 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 11 | 7 | 7
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1 | 3
Investigations (Investigations) | 31 | 19 | 5 | 15
Injury and Complications (Injury, poisoning and procedural complications) | 41 | 38 | 14 | 19
Abdominal Pain (Gastrointestinal disorders) | 2 | 3 | 2 | 2
Injection Site erythema (General disorders) | 2 | 3 | 2 | 3
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 3
Metabolism and Nutritional Disorders (Metabolism and nutrition disorders) | 21 | 14 | 4 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other